CLINICAL TRIAL: NCT01032512
Title: Preoperative Nutrition Support in Major Oncologic Surgery
Brief Title: Clinical Benefits of Preoperative Nutrition Support With Enteral Immune-enhancing Formulas in Surgical Oncology
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: impossibility to include patients in the study
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, MARIA PIA DE LA MAZA, Mrs, University of Chile
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FALP001
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: CANCER
Keywords: IMMUNE-ENHANCING; GLUTAMINE; ARGININE; OMEGA 3 FATTY ACIDS; ONCOLOGIC SURGERY; PREOPERATIVE NUTRITION
MeSH Terms: conditions — Neoplasms | interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMMUNE-ENHANCING (Experimental): 40 patients will be instructed to consume 600 ml of the special "immune-enhancing" formula plus 20 g glutamine (Supportan R + Glutamine plus R, which contain 900 Kcal and 60 g protein/day, with 24.4 g glutamine, 2,2 g arginine and 4.4 g of omega 3 fatty acids, in a lower volume due to its higher energy density).
  Interventions: Dietary Supplement: SUPPORTAN + GLUTAMINE PLUS
- CONTROL (Sham Comparator): 40 patients that do not agree to participate, do not have enough time before the operation, do not tolerate the product and/or drink less than 100 cc/day.
  Interventions: Dietary Supplement: NO PREOPERATIVE NUTRITION SUPPORT

INTERVENTIONS:
Dietary Supplement: SUPPORTAN + GLUTAMINE PLUS — 600 ML OF AN ENERGY DENSE DRINK PLUS 20 G GLUTAMINE POWDER (to give 900 Kcal and 80 g protein/day)
  Other Names: SUPPORTAN
  Arms: IMMUNE-ENHANCING
Dietary Supplement: NO PREOPERATIVE NUTRITION SUPPORT — Patients will be assessed and followed, but will receive no special nutritional support before the surgical procedure
  Other Names: CONTROL
  Arms: CONTROL

SUMMARY:
After surgical treatment, numerous trials using early postoperative enteral or parenteral nutritional support have been attempted, in order to reduce morbidity and mortality. Although it is difficult to compare among heterogeneous interventions, most of them have not been successful, a fact generally attributed to the timing of the intervention. On the other hand, nutrients that become "conditionally essential" under certain stressful circumstances, the so called nutraceuticals, have been incorporated into nutritional formulations. Both facts have prompted the idea of pre or perioperative nutrition support, using specific formulations called "immune enhancing" formulas, containing arginine, nucleotides, glutamine and omega3 fatty acids in varying concentrations. The provision of these nutraceuticals prior and early after the surgical, and particularly in oncologic surgery, theoretically permits to obtain adequate circulating and tissue concentrations for the moment when they are most needed. Exclusive postoperative provision of these substances would not be able to replenish depots and provide them for an adequate immune response and wound healing after surgery. However, regarding the preoperative approach, it is still not know which patients benefit more (less or more severely malnourished), which specific nutrient(s) are responsible for the positive effects, and the precise timing these nutrients should be provided. The present study aims to demonstrate that immune-enhancing formulas are superior to standard enteral products in reducing postoperative nutrition-related complications.

DETAILED DESCRIPTION:
HYPOTHESIS:

Patients receiving enteral nutrition support with immune-enhancing formulas (containing higher concentrations of arginine, glutamine and omega 3 fatty acids compared with standard polymeric formulas) during 7 days before a major oncological surgical procedure, have a lower incidence of nutritional-related postoperative complications, compared with patients without preoperative nutritional supplementation or those supplemented with standard formulas.

OBJECTIVES:

* To put in practice a routine nutritional assessment for every patient that is going to be submitted to major digestive oncologic surgery
* In these patients evaluate adherence and tolerance of enteral drinks, comparing immune-enhancing with the standard polymeric formulations, during 7 days prior to surgery
* To compare frequency of postoperative nutrition-related complications (infections, anastomotic leaks and hospital length of stay), among non-supplemented patients and those receiving preoperative immune-enhancing or standard polymeric formulas.

PATIENTS AND METHODS:

Every patient proposed for major elective digestive oncologic surgery will be invited to a nutritional assessment. Exclusion criteria will be emergency surgery or renal failure (serum creatinine over 1.5 mg/dL). Some patients will not accept or will not be able to attend for several reasons, however they will be assessed by the clinical nutritionist the day of admission, before entering the OR, and followed as the other study patients, and will be considered the control group. Nutritional assessment will include clinical story, dietary recall, Global Subjective Assessment (GSA), calculation of percent weight loss respect habitual weight, anthropometric measurements (height, weight, body mass index) and hand grip strength. Functional involvement will be studied by the Karnofsky score. Among laboratory analysis total proteins, albumin, creatinine, BUN and blood cells for lymphocyte count will be included. All data will be registered in a special chart and then emptied in a computational data base.

After the nutritional assessment, both well nourished and undernourished patients will be instructed to consume an enteral drink, orally or by gastrostomy or enteral feeding tube, during 7 days before surgery. Seventy patients will receive 1 lt per day of a standard polymeric formula (Fresubin 22%, which gives 1000 Kcal and 35 g protein, does not contain free aminoacid nor omega fatty acids, and contains glutamine and arginine concentrations of milk proteins. In order to increase protein intake, 50 g /día of Proteinex R will be added in this group). The other 70 patients will be instructed to consume 600 ml of the special immune-enhancing formula plus 20 g glutamine (Supportan R + Glutamine plus R , which contain 900 Kcal and 60 g protein/day, with 24.4 g glutamine, 2,2 g arginine and 4.4 g of omega 3 fatty acids, in a lower volume due to its higher energy density). Both products are enriched with essential vitamins and minerals. The enteral formulas will be assigned through randomized computer-generated numbers, in an open way. Patients that do not agree to participate, do not have enough time before the operation, do not tolerate the product and drink less than 100 cc/day will be considered control subjects. The enteral products will be sold to the patients directly at the oncologic clinic, both the same prize, and lower to marketing prizes, due to the participation of Fresenius-Kabi in the protocol. However if the patients does not have the means, will receive it for free. All patients will be instructed to maintain their previous diet, adding the enteral supplement, or completing their requirement by tube feeding with standard or specific formulations (e.g. diabetic formulation).

All patients will be followed during the entire postoperative period, registering days of stay at the critical ward, time of mechanical ventilation, days of fever, infections (wound, intra-abdominal, pulmonary, urinary, etc), anastomotic leaks and time of hospitalization.

The participation of Fresenius-Kabi will consist of:

* Paying the enteral formulas, thus avoiding payment for patients (considering that Fundación Arturo Lopez Perez is a private institution, where patients must pay for their treatment, according to their health insurance, which usually exclude nutritional products).
* Collaboration with data registry (nutritional assessment, adherence to the supplements, postoperative complications, etc.) due to the incorporation of one of their professionals (nutritionist) to the study.

ELIGIBILITY:
Inclusion Criteria:

* Every patient submitted for major digestive oncologic surgery in the next 8 to 10 days
* Agrees to participate
* Tolerates formula

Exclusion Criteria:

* Emergency surgery
* Time for surgery less than 8 days
* Serum creatinine > 1.5 mg/dL

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
LENGTH OF HOSPITALIZATION | 30 DAYS

SECONDARY OUTCOMES:
POST OPERATIVE COMPLICATIONS | 60 DAYS
  Registration of all eventual surgical complication after oncologic surgery, both during hospital stay and after 30 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: María Pía de la Maza, M.D., Principal Investigator — INTA, University of Chile; Daniel C. Bunout, M.D., Study Chair — INTA, University of Chile
Locations (1):
- Oncologic Hospital Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] August DA, Huhmann MB; American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.) Board of Directors. A.S.P.E.N. clinical guidelines: nutrition support therapy during adult anticancer treatment and in hematopoietic cell transplantation. JPEN J Parenter Enteral Nutr. 2009 Sep-Oct;33(5):472-500. doi: 10.1177/0148607109341804. No abstract available. PMID 19713551